CLINICAL TRIAL: NCT02540369
Title: PEGASUS: A Prospective obsErvational Study in Patients With Wet aGe-related Macular Degeneration or Diabetic Macular Edema to ASsess the Use of Intravitreal Aflibercept in roUtine Clinical practiceS in Canada
Brief Title: To Describe the Use of Intravitreal Aflibercept and to Describe Follow-up as Well as Treatment Patterns in Patients With Wet Age-related Macular Degeneration (wAMD) or Diabetic Macular Edema (DME) in Routine Clinical Practice in Canada.
Acronym: PEGASUS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 17995
Record Dates: First submitted 2015-08-05; First posted 2015-09-03 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Wet Macular Degeneration
Keywords: Diabetic macular edema; Wet Age-related macular degeneration
MeSH Terms: conditions — Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BAY86-5321- with wAMD: Patients with wet Age Related Macular Degeneration (wAMD) both naïve and previously treated patients
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- BAY86-5321 - with DME: Patients with Diabetic Macular Edema (DME) both naïve and previously treated patients
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Administration by intravitreal injection.Muti-target Anti-VEGF agent. Dosing would be at physicians discretion.

SUMMARY:
To describe the use of intravitreal aflibercept in routine clinical practice and to describe follow-up as well as treatment patterns in patients with wAMD or DME in routine clinical practice in Canada for a study population of treatment naive patients and those who have received prior therapy (anti-VEGF injections, laser, steroids, etc).

ELIGIBILITY:
Inclusion Criteria:

* Age: >= 18 years of age
* Male or female
* Patients with wet AMD (wet age-related macular degeneration) or Diabetic macular edema (DME) who will be treated by intravitreal aflibercept according to the Canadian Product monograph recommendations and routine clinical practice.
* Decision to treat with intravitreal aflibercept prior to patient enrolment as per the physician's routine clinical practice.

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice.
* Patients currently being treated with intravitreal aflibercept. This study will only include patients new to intravitreal aflibercept, both naïve and previously treated with other anti-VEGF therapies.
* Patients who are hypersensitive to this drug, to any ingredient in the formulation, or to any component of the container.
* Patients who are hypersensitive to this drug, to any ingredient in the formulation, or to any component of the container.
* Ocular or peri-ocular infection
* Active intraocular inflammation
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Any concomitant therapy with another agent to treat wet AMD or DME in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wAMD (wet age-related macular degeneration) and DME (Diabetic macular edema) treated by retina specialist/ophthalmologist in selected Canadian clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 2150 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Mean change of visual acuity. | Baseline and 12 months
  Treatment in naïve and previously treated patients for wAMD and DME.

SECONDARY OUTCOMES:
Change of visual acuity. | Baseline and 12 months
  For the overall population
Change of visual acuity by number of Injections. | Baseline and 12 months
  In 2 sub groups
Change in Retinal thickness. | Baseline and 12 months
Treatment patterns used in routine clinical practice setting. | Up to 12 months
  Number of visits and examinations per patient
Maximum interval between treatments. | Up to 12 months
Mean time between injections. | Up to 12 months
Number of injections at 12 months. | Up to 12 months
Time to achieve stability of disease. | Up to 12 months
Number of injections in a year to achieve stability of disease. | Up to 12 months
In previously treated subpopulation duration of previous treatments | At Baseline
In previously treated subpopulation type of previous treatments. | At Baseline
In previously treated subpopulation reason to switch to Eylea. | At Baseline
  Some of the reasons are recurrence of fluid, new hemorrhage - bleed, decreased vision, lack of compliance, patient request, etc.
Proportion of patients with no fluid determined by Optical coherence tomography (OCT). | At 4 months, At 12 months
  Absence of fluid would be determined by physician's judgment in the AMD population.
Numbers of patients require adjunctive therapies. | Up to 12 months
  For Diabetic macular edema patients
Type of adjunctive therapies required by patients | Up to 12 months
  For Diabetic macular edema patients adjunctive therapies as focal laser, steroids, etc.
Number of participants with adverse events as a measure of safety and tolerability. | Up to 12 months
Presence of pigment epithelial detachment (PED) (Y/N) | Baseline and at 12 months
  For Age-related macular degeneration patients.
Diabetic retinopathy severity (mild, moderate, severe). | Up to 12 months
  For Diabetic macular edema patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Canada